CLINICAL TRIAL: NCT07319845
Title: A Phase 2, Multicenter, Open-Label, Single-arm Study to Evaluate the Efficacy and Safety of TAK-226 for Transfusion-Dependent Anemia in Japanese Patients With Very Low, Low, or Intermediate Risk Myelodysplastic Syndromes
Brief Title: A Study of TAK-226 for Transfusion-Dependent Anemia in Japanese Patients With Lower-Risk Myelodysplastic Syndromes
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAK-226-2001
Record Dates: First submitted 2025-12-22; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Myelodysplastic Syndromes
Keywords: Drug Therapy
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TAK-226 (Experimental): Participants will receive the study drug, TAK-226, administered subcutaneously every four weeks (Q4W), up to 48 weeks or until the end of for approximately one year during Treatment Period.
  Interventions: Drug: TAK-226

INTERVENTIONS:
Drug: TAK-226 — TAK-226 subcutaneous injection
  Other Names: Elritercept; KER-050

SUMMARY:
The main aim of the study is to evaluate how TAK-226 improves symptoms of transfusion-dependent anemia in Japanese patients with lower-risk myelodysplastic syndromes.

The study consists of Screening Period (up to 6 weeks), Treatment Period , Safety Follow-Up Period (8 weeks), and Long-Term Follow-Up Period (5 years from the first dose of the study drug or 3 years after the last dose, whichever is longer).

Participants of this study will be administered TAK-226 during Treatment Period. Subsequently, the participants will be monitored for side effects related to the study treatment during Safety Follow-Up Period and Long-Term Follow-Up Period. The approximate duration of participation for a participant is up to approximately 6 years.

During the study period, participants will visit the study clinic/hospital multiple times as per the study schedule. During Treatment Period, the participants will come to the clinic/hospital approximately every two to four weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Participants or their legally authorized representative must be willing and able to sign the ICF and to adhere to the protocol requirements.
2. Japanese adult male or female participant ≥18 years of age at the time of signing informed consent.
3. Diagnosis of MDS with or without RS (as determined in an evaluable bone marrow aspirate collected at Screening to confirm diagnosis) according to WHO 2016 classification that meets the IPSS-R classification of very low-, low-, or intermediate-risk MDS.

   Note: Due to expected impacts of transfusion, Hgb values from blood samples collected within 14 days following an RBC transfusion and platelet count obtained within 7 days following a platelet transfusion cannot be used to evaluate IPSS-R for eligibility.
4. Transfusion dependence assessed in the 16 weeks immediately preceding enrollment in two 8-week blocks classified as either:

   a. LTB, defined as 4 to 7 RBC units per 16 weeks; or b. HTB, defined as ≥8 RBC units per 16 weeks; and c. For all participants: i. Only transfusion events for a pretransfusion Hgb <10 g/dL are counted toward eligibility; ii. At least 1 transfusion event in each 8-week block and a minimum of 2 transfusion events separated by ≥7 days within the 16-week period immediately preceding enrollment; and iii. No consecutive 56-day period can be RBC transfusion-free during the 16 week period immediately preceding enrollment.

   Note: Only transfusions for the disease under study will be counted towards classification for LTB or HTB participants. Transfusions for intercurrent diseases (bleeding, surgical procedure, infection, etc.) are not considered.
5. Refractory or intolerant to prior ESA treatment (discontinued ≥4 weeks before enrollment), or unlikely to respond to ESA treatment, defined as follows:

   a. Refractory to prior ESA treatment: documentation of nonresponse or a response that was no longer maintained with a prior ESA-containing regimen, either as a single agent or combination (eg, with granulocyte colony-stimulating factor [G-CSF]); ESA regimen must have been either: i. Recombinant human EPO ≥40,000 IU/week for ≥8 doses or equivalent; or ii. Darbepoetin alpha ≥500 mcrg every 3 weeks for ≥4 doses or equivalent. b. Intolerant to prior ESA treatment: documentation of discontinuation of a prior ESA containing regimen, either as a single agent or combination (eg, with G-CSF), at any time after introduction due to intolerance or an AE.

   c. Unlikely to respond to ESA treatment: low chance of response to ESA based on an endogenous serum EPO level >200 U/L.

   Note: Due to expected impacts of transfusion on EPO levels, blood samples collected within the 14 days following an RBC transfusion or within 7 days following a platelet transfusion cannot be used to evaluate serum EPO level for eligibility.
6. Less than 5% blasts in an evaluable bone marrow aspirate collected at Screening.
7. ECOG performance status of 0 to 2.
8. Women of childbearing potential (WOCBP), defined as a sexually mature woman who has not undergone surgical sterilization or who has not been naturally postmenopausal for at least 12 consecutive months must

   1. Agree to use 1 highly effective method of contraception and 1 additional effective (barrier) method at the same time, from the time of signing the informed consent through 60 days after the last dose of study drug; or
   2. Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the participant. (Periodic abstinence [eg, calendar, ovulation, symptothermal, postovulation methods], withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception.)
9. Male participants must, even if he is surgically sterilized (ie, status postvasectomy),

   1. Agree to practice effective barrier contraception the time of signing the informed consent through 60 days after the last dose of study drug; or
   2. Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the participant. (Periodic abstinence [eg, calendar, ovulation, symptothermal, postovulation methods], withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception.)

Exclusion Criteria:

Medical History

1. Del(5q) MDS or therapy-related (secondary) MDS.
2. Anemia due to any other known cause (eg, thalassemia, hemolytic anemia, bleeding events, or deficiency of iron, B12, and/or folate).
3. Receipt of RBC transfusion for any reason(s) other than underlying MDS within 16 weeks before enrollment.
4. Clinically significant cardiovascular disease defined as:

   1. New York Heart Association heart disease class III or IV;
   2. Fridericia corrected QT (QTcF) interval >500 milliseconds during Screening;
   3. Presence of uncontrolled hypertension defined as mean systolic blood pressure ≥160 mm Hg or diastolic blood pressure ≥100 mm Hg during Screening; or
   4. Uncontrolled arrhythmia, myocardial infarction, or unstable angina within 6 months before Screening.
5. Known ejection fraction <35%, confirmed by a local echocardiogram performed during Screening, or a previously performed echocardiogram if collected within 6 months before Screening.
6. Stroke, deep vein thrombosis, or pulmonary embolism within 6 months before Screening.
7. Any known history of acute myeloid leukemia (AML).
8. Prior history of malignancies, other than MDS, unless the participant has been free of the disease (including completion of any treatment, including maintenance, for prior malignancy) for ≥5 years. However, participants with a history or concurrent diagnosis of the following conditions are allowed if not requiring systemic therapy:

   1. Basal or squamous cell carcinoma of the skin;
   2. Carcinoma in situ of the cervix;
   3. Carcinoma in situ of the breast; and/or
   4. Incidental histologic finding of prostate cancer (T1a or T1b using the tumor, node, metastasis [TNM] clinical staging system).
9. History of solid organ or bone marrow transplantation.
10. Active infection requiring intravenous antibiotics within 28 days or oral antibiotics within 14 days before enrollment.
11. History of or known active or chronic infection with HIV, active infectious hepatitis B virus (HBV), or active infectious hepatitis C virus (HCV). Participants who are positive for hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), or hepatitis B surface antibody (HBsAb) may be eligible for enrollment if their hepatitis B viral load is below the limit of detection. Participants who are positive for hepatitis C virus antibodies (HCVAb) may be enrolled if their hepatitis C viral load is below the limit of detection.
12. Body mass index ≥40 kg/m^2.
13. Major surgery within 28 days before enrollment.
14. History of allergy/anaphylaxis to investigational medicinal product (IMP) excipients (refer to the current elritercept [TAK 226] IB for a list of excipients) or recombinant proteins.

    Treatment History
15. Prior use of TAK 226, luspatercept, imetelstat, or sotatercept.
16. Prior use of hypomethylating agents (HMAs), isocitrate dehydrogenase inhibitor, lenalidomide, or immunosuppressive therapy given for treatment of MDS.
17. Iron chelation therapy initiated within 8 weeks before enrollment. Participants on stable doses of iron chelation therapy for ≥8 weeks are allowed.
18. Vitamin B12 or folate therapy initiated within 4 weeks before enrollment. Participants on stable replacement doses for ≥4 weeks and without ongoing concurrent vitamin B12 or folate deficiency are allowed.
19. Androgen use within 8 weeks before enrollment. Participants on stable androgen dosing for hypogonadism for ≥8 weeks are allowed.
20. High-dose corticosteroid use within 4 weeks before enrollment. Participants on stable chronic steroid doses of prednisone/prednisolone ≤10 mg/day or corticosteroid equivalent for ≥4 weeks are allowed.
21. Treatment with any investigational drug within 28 days before Screening or, if the half-life of the product is known, within 5 times the half-life before Screening, whichever is longer.
22. Ongoing participation in another interventional clinical study. Laboratory Exclusions (during Screening)
23. Serum EPO level >500 U/L. Note: Due to expected impacts of transfusion on EPO levels, laboratory results from blood samples collected within the 14 days following an RBC transfusion cannot be used to evaluate serum EPO level for eligibility.
24. Platelet count ≥450×10^3/mcrL or ≤25×10^3/mcrL. Note: Due to expected impacts of transfusion, laboratory results from blood samples collected within the 7 days following a platelet transfusion cannot be used to evaluate platelet count for eligibility.
25. Absolute neutrophil count ≤500/mcrL
26. Serum AST or ALT ≥3×the upper limit of normal (ULN).
27. Total bilirubin ≥2×ULN unless attributable to Gilbert syndrome.
28. Ferritin ≤50 mcrg/L.
29. Folate ≤2.0 ng/mL.
30. Vitamin B12 ≤200 pg/mL.
31. Estimated glomerular filtration rate <30 mL/min/1.73m^2 as determined by Japanese Society of Nephrology. Calculated by the correction formula for Japanese.

    eGFR=194× (serum creatinine value)^-1.094× (age)^-0.287× (sex correction factor), Sex correction factor: 0.739 in female.

    Miscellaneous
32. Pregnant or lactating female. Note: Participants who may be in the very early stage of pregnancy based on the doctor's interview with a negative pregnancy test are excluded from the study. Participants who are lactating will be eligible if they discontinue breastfeeding from before the first dose of study drug until 60 days after the last dose of study drug.
33. Any other condition not specifically noted above that, in the opinion of the investigator, would preclude the participant from participating in the study or could confound interpretation of data from the study.
34. Investigational site staff members directly involved in the conduct of the study and site staff members otherwise supervised by the investigator, employees of the Sponsor or contract research organization (CRO) directly involved in the conduct of the study, or immediate family members (defined as a spouse, parent, child, or sibling, whether biological or legally adopted).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2026-02-06 (Estimated); Primary Completion 2028-06-26 (Estimated); Study Completion 2033-01-10 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Transfusion Independence (TI) for Greater Than or Equal to 8 Weeks from Baseline through Week 24 | Baseline, Up to Week 24
  Transfusion independence is defined as the absence of any red blood cells (RBC) transfusions in a period of at least 8 weeks after the first dose of the study treatment through week 24.

SECONDARY OUTCOMES:
Percentage of Participants Achieving TI for Greater Than or Equal to 24 Weeks from Baseline through Week 48 | Baseline, Up to Week 48
  Transfusion independence is defined as the absence of any red blood cells (RBC) transfusions in a period of at least 24 weeks after the first dose of the study treatment through week 48.
Percentage of Participants with High Transfusion Burden (HTB) Achieving TI for Greater Than or Equal to 8 Weeks from Baseline through Week 24 | Baseline, Up to Week 24
  Transfusion independence is defined as the absence of any red blood cells (RBC) transfusions in a period of at least 8 weeks after the first dose of the study treatment through week 24.
Percentage of Participants Achieving Mean Haemoglobin (Hgb) Increase of Greater Than or Equal to 1.5 grams per deciliter (g/dL) for Greater Than or Equal to 8 Weeks from Baseline through Week 24 | Baseline, Up to Week 24
Number of Participants with Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | Up to approximately 6 years
  An AE is any untoward medical occurrence in a clinical trial participant, temporally associated with the use of the trial intervention, whether or not the occurrence is considered related to the trial intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of the trial intervention. A TEAE is defined as an AE that commences on or after the first dose of the study treatment and within 60 days after the last dose of the study treatment, or analysis cutoff date, whichever is earlier. An SAE is any untoward medical occurrence that, at any dose: results in death, is life threatening, requires in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a medically important event.
Change from Baseline in Clinical Laboratory Values, Vital Signs, and Electrocardiograms (ECGs) | From the time of signing the informed consent form through safety follow-up, approximately 16 months
  Change from baseline in clinical laboratory values, vital signs, and ECGs will be assessed.
Serum Concentration of TAK-226 | Baseline, and multiple time points up to the end of Treatment Period (approximately 12 months)
  TAK-226 time-concentration data will be assessed.
Number of Participants with Treatment-Emergent Anti-Drug Antibody (ADA) | Up to the end of Safety Follow-Up Period (approximately 4 months)
ADA Titer | Baseline, and multiple time points up to approximately 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/